CLINICAL TRIAL: NCT03316586
Title: A Phase II Study of Nivolumab in Combination With Cabozantinib for Metastatic Triple-negative Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Bristol-Myers Squibb (Industry); Exelixis (Industry)
Responsible Party: Principal Investigator, Sara Tolaney, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-324
Record Dates: First submitted 2017-10-18; First posted 2017-10-20 (Actual); Results first posted 2021-12-28 (Actual); Last update posted 2021-12-28 (Actual); Status verified 2021-11

CONDITIONS: Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Nivolumab; cabozantinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nivolumab + Cabozantinib (Experimental): * Nivolumab was administered every 28 days at a dose of 480mg given intravenously over 30 minutes (+/- 10 minutes) using a volumetric pump with 0.2 to 1.2 micron pore size, low protein binding polyethersulfone membrane in-line filter
  * Cabozantinib was administered orally, once daily for 28 days at a dose of 40 mg.
  Interventions: Drug: Nivolumab; Drug: Cabozantinib

INTERVENTIONS:
Drug: Nivolumab — Nivolumab is an experimental antibody drug that may make the immune response more active against cancer.
  Other Names: Opdivo
Drug: Cabozantinib — Cabozantinib may help to shrink or stabilize breast cancer
  Other Names: Cabometyx

SUMMARY:
This research study is studying a combination of drugs as a possible treatment for metastatic triple-negative breast cancer.

The drugs involved in this study are:

* Cabozantinib (XL184)
* Nivolumab

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational intervention to learn whether the intervention works in treating a specific disease. "Investigational" means that the intervention is being studied.

The FDA (the U.S. Food and Drug Administration) has not approved the combination of Nivolumab and Cabozantinib as a treatment for any disease.

The FDA has not approved Cabozantinib for this specific disease but it has been approved for other uses. The FDA (the U.S. Food and Drug Administration) has not approved nivolumab for this specific disease but it has been approved for other uses.

Cabozantinib has been used in some phase I studies and information from those other research studies suggests that cabozantinib may help to shrink or stabilize breast cancer.

Cancers are recognized by the immune system, and under some circumstances, the immune system may control or even eliminate tumors. An antibody is a natural protein made by the immune system that binds other proteins and molecules to fight infection and its ill effects. Antibodies stimulating the immune system have been developed for treatment of human cancers. Nivolumab is an experimental antibody drug that may make the immune response more active against cancer.

In this research study, the investigators are looking at how the participant's type of breast cancer responds to the combination of cabozantinib and nivolumab.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically or cytologically confirmed invasive breast cancer, with metastatic disease. Participants without pathologic or cytologic confirmation of metastatic disease should have unequivocal evidence of metastasis from physical examination or radiologic evaluation.
* Estrogen-receptor and progesterone-receptor expression both <10% by immunohistochemistry (IHC) and human epidermal growth factor receptor 2 (HER2) negative by IHC or non-amplified as determined by the current American Society of Clinical Oncology (ASCO)/CAP (College of American Pathologists) criteria. If patient has more than one histological result, the most recent one has to be considered for inclusion.
* Participants must have measurable disease by RECIST version 1.1
* Participants must agree to undergo a research biopsy, if tumor is safely accessible, at baseline and 7-14 days prior to Cycle 3 Day 1. Participants for whom newly-obtained samples cannot be provided (e.g. inaccessible or participant safety concern) may submit an archived specimen.

Note: After the first 6 participants undergo biopsy on cabozantinib, we will review their adverse event profiles to ensure no more than a 20% rate of grade 3 or higher bleeding or wound healing complications occur. If more than 2 patients (>20%) have safety concerns, we will reassess the safety of collecting the research biopsies. Full review of all grade (including grade 1 and 2) may also prompt changes and will be reviewed by the study team. Exelixis may be consulted if necessary.

* Prior chemotherapy: Participants may have received 0-3 prior chemotherapeutic regimens for metastatic breast cancer and must have been off treatment with chemotherapy for at least 14 days prior to registration. Participants should also be adequately recovered from acute toxicities of prior treatment.
* Prior biologic therapy: Patients must have discontinued all biologic therapy at least 14 days prior to registration.
* Prior radiation therapy: Patients may have received prior radiation therapy in either the metastatic or early-stage setting. Radiation therapy must be completed per the following timelines:

  * Radiotherapy to the thoracic cavity or abdomen within 4 weeks prior to registration.
  * Radiotherapy to bone lesions within 2 weeks prior to registration.
  * Radiotherapy to any other site within 4 weeks prior to registration.
* In all cases, there must be complete recovery and no ongoing complications from prior radiotherapy.
* The subject is ≥18 years old.
* ECOG (Eastern Cooperative Oncology Group) performance status ≤1(Karnofsky ≥60%, see Appendix A)
* Participants must have normal organ and marrow function as defined below:

  * absolute neutrophil count ≥1,000/microliter (mcL)
  * platelets ≥100,000/mcL
  * hemoglobin ≥ 9 g/dl
  * total bilirubin ≤1.5 × institutional upper limit of normal (ULN) (or 2.0 x ULN in patients with documented Gilbert's Syndrome)
  * Aspartate aminotransferase (AST) / Alanine transaminase (ALT) ≤2.5 × institutional ULN or ≤ 3 × institutional ULN for participants with documented liver metastases
  * creatinine <1.5 ×institutional ULN OR creatinine clearance ≥40 mL/min (using Cockcroft-Gault formula) for participants with creatinine levels above institutional ULN.
  * Urine protein/creatinine ratio (UPCR) ≤1
* Female subjects of childbearing potential must have a negative pregnancy test at screening
* Childbearing potential is defined as: participants who have not reached a postmenopausal state (≥ 12 continuous months of amenorrhea with no identified cause other than menopause) and has not undergone surgical sterilization (removal of ovaries and/or uterus).
* Female and male participants of childbearing potential must agree to use an adequate method of contraception. Contraception is required starting with the first dose of study medication through 150 days (5 months) after the last dose of study medication . Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, established and proper use of hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.
* Participants on bisphosphonates may continue receiving bisphosphonate therapy during study treatment.
* The participant is capable of understanding and complying with the protocol and has signed the informed consent document

Exclusion Criteria:

* Major surgery within 12 weeks before the first dose of study treatment. Complete wound healing from major surgery must have occurred 1 month before the first dose of study treatment. Minor surgery (including uncomplicated tooth extractions) within 28 days before the first dose of study treatment with complete wound healing at least 10 days before the first dose of study treatment. No clinically relevant ongoing complications from prior surgery are not eligible.
* The participant has tumor in contact with, invading, or encasing major blood vessels or radiographic evidence of significant cavitary pulmonary lesions.
* The subject has pathologic evidence of tumor invading the GI tract (esophagus, stomach, small or large bowel, rectum or anus), or any evidence of endotracheal or endobronchial tumor within 28 days before the first dose of cabozantinib;
* Concurrent administration of other anti-cancer therapy within 14 days of starting protocol therapy and during the course of this study.
* The participant has received another investigational agent within 14 days of the first dose of study drug.
* The participant has received a prior c-Met inhibitor
* Has received prior therapy with an anti-programmed cell death-1 (PD-1), anti-PD-L1, anti-PD-L2, anti-CD137, or anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including pembrolizumab, ipilimumab, and any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways)
* Known brain metastases that are untreated, symptomatic, or require therapy to control symptoms. Participants with a history of treated central nervous system (CNS) metastases are eligible. Treated brain metastases are defined as those having no evidence of progression for ≥ 1 month after treatment, and no ongoing requirement for corticosteroids, as ascertained by clinical examination and brain imaging (magnetic resonance imaging or CT scan) completed during screening. Any corticosteroid use for brain metastases must have been discontinued without the subsequent appearance of symptoms for ≥2 weeks prior to registration. Treatment for brain metastases may include whole brain radiotherapy, radiosurgery, or a combination as deemed appropriate by the treating physician. Participants with CNS metastases treated by neurosurgical resection or brain biopsy performed within 2 months before day 1 will be excluded.
* The subject has uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

  * Cardiovascular disorders including:
  * Congestive heart failure (CHF): New York Heart Association (NYHA) Class III (moderate) or Class IV (severe) at the time of screening;
  * Concurrent uncontrolled hypertension defined as sustained blood pressure (BP) > 150 mm Hg systolic or > 100 mm Hg diastolic despite optimal antihypertensive treatment within 7 days of the first dose of study treatment;
  * Any history of congenital long QT syndrome;
  * Any of the following within 6 months before the first dose of study treatment:
  * unstable angina pectoris;
  * clinically-significant cardiac arrhythmias;
  * stroke (including transient ischemic attack (TIA), or other ischemic event);
  * myocardial infarction;
  * GI disorders particularly those associated with a high risk of perforation or fistula formation including:
  * Tumors invading the GI tract, active peptic ulcer disease, active inflammatory bowel disease (eg, Crohn's disease), active diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, acute pancreatitis or acute obstruction of the pancreatic duct or common bile duct, or gastric outlet obstruction
  * Abdominal fistula, GI perforation, bowel obstruction, intra-abdominal abscess within 6 months before randomization, Note: Complete healing of an intra-abdominal abscess must be confirmed prior to randomization
* Other clinically significant disorders that would preclude safe study participation;
* Corrected Fridericia's QT interval (QTcF) interval >500 msec Note: Three ECGs must be performed for eligibility determination. If the average of these three consecutive results for QTcF is ≤ 500 msec, the subject meets eligibility in this regard.
* Thromboembolic events requiring therapeutic anticoagulation. Concomitant anticoagulation with oral anticoagulants (eg, warfarin, direct thrombin and Factor Xa inhibitors), platelet inhibitors (eg, clopidogrel) are prohibited.

Note: Low-dose aspirin for cardioprotection (per local applicable guidelines) and low-dose low molecular weight heparin (LMWH) are permitted (in subjects who are on a stable dose of LMWH for at least 6 weeks before the first dose of study treatment, and who have had no clinically significant hemorrhagic complications from the anticoagulation regimen or the tumor).

Note: Subjects with a venous filter (eg vena cava filter) are not eligible for this study).

* Individuals with a history of different malignancy are ineligible except for the following circumstances. Individuals with a history of other malignancies are eligible if they have been disease-free for at least 3 years or are deemed by the investigator to be at low risk for recurrence of that malignancy.
* Participant has an active infection requiring IV antibiotics
* Patient has a medical condition that requires chronic systemic steroid therapy or on any other form of immunosuppressive medication. For example, participants with autoimmune disease that requires systemic steroids or immunosuppression agents should be excluded. Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* The participant is known to be positive for the human immunodeficiency virus (HIV), HepBsAg, or Hepatitis C virus (HCV) RNA. HIV-positive participants on combination antiretroviral therapy are ineligible.
* Known hypersensitivity to any of the components of cabozantinib or nivolumab.
* The participant has received a live vaccine within 28 days prior to the first dose of trial treatment and while participating in the trial. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster, yellow fever, rabies, bacille Calmette-Guerin (BCG), and typhoid vaccine. The use of the inactivated seasonal influenza vaccine (Fluzone®) is allowed.
* The subject has experienced any of the following:

  * Clinically significant gastrointestinal bleeding within 6 months before the first dose of study treatment
  * Clinically significant hemoptysis within 3 months of the first dose of study treatment
  * Any other signs indicative of pulmonary hemorrhage within 3 months before the start of study treatment
* The participant is unable to swallow oral dosage forms.
* The participant is pregnant or breastfeeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-11-30 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sara Tolaney, MD, MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Nivolumab + Cabozantinib: * Nivolumab was administered every 28 days at a dose of 480mg given intravenously over 30 minutes (+/- 10 minutes) using a volumetric pump with 0.2 to 1.2 micron pore size, low protein binding polyethersulfone membrane in-line filter
  * Cabozantinib was administered orally, once daily for 28 days at a dose of 40 mg.
  Nivolumab: Nivolumab is an experimental antibody drug that may make the immune response more active against cancer.
  Cabozantinib: Cabozantinib may help to shrink or stabilize breast cancer
Period: Overall Study
Arm/Group | Nivolumab + Cabozantinib
Started | 18
Completed | 0
Not Completed | 18
Not completed — Adverse Event | 2
Not completed — Physician Decision | 3
Not completed — Lack of Efficacy | 10
Not completed — still on treatment | 1
Not completed — Patient needed radiation therapy | 1
Not completed — Physician Decision to send patient for breast surgery | 1

BASELINE CHARACTERISTICS:
Arm/Group | Nivolumab + Cabozantinib
Number analyzed (Participants) | 18
Age, Continuous [Median (Full Range); unit: years] | 58 [41 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 15
  More than one race | 1
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18
ECOG [Count of Participants; unit: Participants] — The ECOG (Eastern Cooperative Oncology Group) Scale of Performance Status describes a patient's level of functioning in terms of their ability to care for themselves, daily activity, and physical ability (walking, working, etc.). This is a numbering scale of 0 to 5. The higher the number, the worse the performance status. Zero (0) refers to being full active. 5 is dead.
  Participants
    0 | 18
    1 | 0
Stage at initial Diagnosis [Count of Participants; unit: Participants] — The stage of breast cancer is determined by the cancer's characteristics such as how large it is and whether or not it has hormone receptors. This is usually expressed as a number on a scale of 0 through IV, with stage 0 describing non-invasive cancers that remain within their original location and stage IV describing invasive cancers that have spread outside the breast to other parts of the body.
  Participants
    I | 3
    II | 6
    III | 2
    IV | 5
    Unknown | 2
Disease free interval [Count of Participants; unit: Participants] — It is measured from the primary diagnosis to the diagnosis of metastatic cancer.
  Participants
    De novo | 5
    <=2 years | 4
    >2 years | 5
    Date missing | 4
Sites of disease -- lung pleural [Count of Participants; unit: Participants] | 6
Sites of disease -- liver [Count of Participants; unit: Participants] | 7
Sites of disease -- bone [Count of Participants; unit: Participants] | 8
Sites of disease -- Breast/chest wall [Count of Participants; unit: Participants] | 7
Sites of disease -- Lymph node [Count of Participants; unit: Participants] | 11
Sites of disease -- Soft tissue [Count of Participants; unit: Participants] | 3
Adjuvant or neoadjuvant hormonal therapy [Count of Participants; unit: Participants] | 1
Adjuvant or or neoadjuvant anthracycline [Count of Participants; unit: Participants] | 12
Adjuvant or neoadjuvant taxane [Count of Participants; unit: Participants] | 12
Lines of chemotherapy for metastasis or recurrence [Median (Full Range); unit: line] | 1 [0 to 3]
Lines of chemotherapy for metastasis or recurrence [Count of Participants; unit: Participants]
  0 | 5
  1 | 6
  2 | 5
  3 | 2
Prior metastatic chemotherapy -- Anthracycline [Count of Participants; unit: Participants] | 4
Prior metastatic chemotherapy -- Taxane [Count of Participants; unit: Participants] | 5
Prior metastatic chemotherapy -- Platinum [Count of Participants; unit: Participants] | 11
Prior metastatic chemotherapy -- Capecitabine [Count of Participants; unit: Participants] | 2
Prior metastatic chemotherapy -- Eribulin [Count of Participants; unit: Participants] | 2
Prior metastatic chemotherapy -- Other chemotherapy [Count of Participants; unit: Participants] | 6
ER, PR, and HER2 status at study entry [Count of Participants; unit: Participants] — ER: Estrogen receptors PR: progesterone receptors
  Participants
    ER and/or PR-positive (≤10%), HER2-negative | 2
    ER and PR negative, HER2-negative | 16
PD-L1 positive cells [Count of Participants; unit: Participants] | 1
TILs in metastatic samples [Count of Participants; unit: Participants] — TILs: tumor-infiltrating lymphocytes
  Participants | 3

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Overall response rate (ORR) is defined as the percentage of patients with complete or partial response evaluated by RECIST 1.1. Per RECIST 1.1: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 2 years
Population: For this Phase II trial, the efficacy evaluable population is a modified intent-to-treat (ITT) population. The modified ITT population consists of all patients who initiate protocol therapy, even if there are major protocol therapy deviations.
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab + Cabozantinib
Number analyzed (Participants) | 18
Participants | 1

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Toxicities will be defined according to NCI CTCAE, Version 4.0
Time Frame: 2 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab + Cabozantinib
Number analyzed (Participants) | 18
Participants | 18

3. Secondary Outcome: Clinical Benefit Rate
Description: Clinical Benefit Rate (CBR) will be determined by looking at the number of subjects who have either a complete response, partial response, or stable disease for greater than or equal to 24 weeks, per RECIST 1.1
Time Frame: 2 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab + Cabozantinib
Number analyzed (Participants) | 18
Participants | 3

4. Secondary Outcome: Progression Free Survival Rate
Description: Progression free survival is defined from the study entry to first documented evidence of disease progression by RECIST 1.1 or death of any cause, whichever occurs first. Patients alive with no progression are censored at the last disease assessment.
Time Frame: 5 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab + Cabozantinib
Number analyzed (Participants) | 18
months | 3.6 [1.9 to 6.9]

5. Secondary Outcome: Overall Response Rate Per Immune Criteria
Description: ORR will be determined according to immune-related response criteria (irRC). Per irRC, irComplete Response (irCR) refers to complete disappearance of all target lesions. irPartial Response (irPR) refers to decrease, relative to baseline, of 50% or greater in the sum of the products of the two largest perpendicular diameters of all target and all new measurable target lesions (i.e., Percentage Change in Tumor Burden). ORR per irRC is irCR + irPR.
Time Frame: 2 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab + Cabozantinib
Number analyzed (Participants) | 18
Participants
  irPR | 1
  irSD | 14
  irPD | 2
  not evaluable | 1

ADVERSE EVENTS:
Time Frame: AE data were collected every cycle from the time of the first dose of the study treatment, through the end of the treatment. Vital status was followed even after patients were off treatment. AEs, including overall mortality, were observed up to 60 months.
Description: Serious AEs (SAE) were defined as events with treatment-attribution of possibly, probably or definitely and grade 3 or higher. All remaining AEs are classified as Other AEs (OAE) including grade 3 or higher events with treatment-attribution of unlikely and unrelated plus all grade 1 and 2 events. Maximum grade toxicity by type was then calculated within SAE and OAE datasets. No further data is available to specify classification of other beyond the general term.
Arm/Group | Nivolumab + Cabozantinib
All-Cause Mortality (participants affected / at risk) | 3/18
Serious Adverse Events (participants affected / at risk) | 13/18
Other Adverse Events (participants affected / at risk) | 17/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab + Cabozantinib (N=18)
Anemia (Blood and lymphatic system disorders) | 1
Endocrine disorders - Other, specify (Endocrine disorders) | 1
Small intestinal perforation (Gastrointestinal disorders) | 1
Edema trunk (General disorders) | 1
Fatigue (General disorders) | 2
Appendicitis (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 3
Dehydration (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Syncope (Nervous system disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 3
Hypertension (Vascular disorders) | 2
Thromboembolic event (Vascular disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab + Cabozantinib (N=18)
Anemia (Blood and lymphatic system disorders) | 1
Lymph node pain (Blood and lymphatic system disorders) | 1
Palpitations (Cardiac disorders) | 1
Endocrine disorders - Other, specify (Endocrine disorders) | 1
Hyperthyroidism (Endocrine disorders) | 3
Hypothyroidism (Endocrine disorders) | 7
Abdominal pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 5
Dry mouth (Gastrointestinal disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 2
Oral pain (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Death NOS (General disorders) | 1
Edema face (General disorders) | 1
Edema limbs (General disorders) | 4
Edema trunk (General disorders) | 1
Fatigue (General disorders) | 7
Pain (General disorders) | 2
Allergic reaction (Immune system disorders) | 1
Infections and infestations - Other, specify (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Upper respiratory infection (Infections and infestations) | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1
Wound complication (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 6
Aspartate aminotransferase increased (Investigations) | 9
Creatinine increased (Investigations) | 1
Neutrophil count decreased (Investigations) | 4
Platelet count decreased (Investigations) | 1
Weight loss (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 7
Dehydration (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 5
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 6
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Dysgeusia (Nervous system disorders) | 4
Headache (Nervous system disorders) | 2
Peripheral sensory neuropathy (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Chronic kidney disease (Renal and urinary disorders) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 4
Alopecia (Skin and subcutaneous tissue disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 2
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 7
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 5
Thromboembolic event (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
Only one of the first 18 patients had a PR. The study therefore did not meet the prespecified criteria to proceed to the second stage of the trial, and it was closed to further accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-09): https://cdn.clinicaltrials.gov/large-docs/86/NCT03316586/Prot_SAP_000.pdf